CLINICAL TRIAL: NCT03437798
Title: Exploring Genomic Determinants of Periodontal Disease Via Shared Genetic Pathways With Cardiovascular Disease, Diabetes, and Bone Density
Brief Title: Genomic Determinants and Shared Genetic Pathways of Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: Brigham and Women's Hospital (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Yau-Hua Yu, Assistant Professor, Tufts University
Other Study IDs: HH1804; 1K23DE026804-01 (NIH)
Record Dates: First submitted 2018-01-02; First posted 2018-02-19 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Periodontal Diseases; Diabetes; Osteoporosis; Cardiovascular Risk Factor
Keywords: Periodontal Disease; Diabetes; Osteoporosis; Cardiovascular Risk Factor; Genomic
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Disease status — Women who reported periodontal disease diagnosis/condition

SUMMARY:
Despite significant improvement in treating periodontal disease (PD) and the identification of multiple risk factors, little is known about the specific contribution of genetics to PD pathogenesis. Several genomewide association studies (GWAS) of PD have been published, but only one reported locus has reached the threshold for genome-wide significance. Epidemiological studies and biological experiments established associations and suggested common pathogenetic pathways between PD and cardiovascular disease (CVD), diabetes (DM), and osteoporosis. The overall objective is to identify genetic loci for PD as a first step toward a better understanding of PD pathogenesis. In a preliminary study in the Women's Genome Health Study (WGHS), new-onset cases of PD were associated with a family history of myocardial infarction (MI). Further preliminary analyses presented shared phenotypic variation of PD/CVD, PD/DM, or PD/osteoporosis that could be accounted by the whole-genome genetic matrices. Several variants from the GWAS catalog of bone density and family history of MI were found correlated with PD in the WGHS. Based on these findings and the literature, the central hypothesis is that there are common pathogenetic links between PD and these other diseases and that GWAS using the comorbidity case definitions will help identify potential common loci.

DETAILED DESCRIPTION:
Three specific aims are proposed to refine and validate the PD status in the Women's Health Study (WHS/WGHS) to improve the phenotypic characterization of GWAS of PD: (1) Addition of CDC-AAP (Centers for Disease Control - American Academy of Periodontology) periodontal disease instrument to the WHS annual follow-up survey. (2) Validate existing Periodontal Disease (PD) status in the WHS/WGHS (subset). Request of dental records for 180 women sampled from the WHS who had reported diagnosis of PD in the past. (3) Correlation and validation analysis of new periodontal disease information with requested dental record (most recently dated). Phone interviews and request of dental records for 180 women sampled from the WHS/WGHS who visited a dentist within recent 36 months.

In addition, the investigators propose to identify genetic determinants of PD shared with CVD, DM, or osteoporosis via an integrative computational biological networks approach. Although the systemic links between PD vs. DM, CVD or osteoporosis have been established in clinical genetics as well as in experimental models, high-throughput investigations for gene-gene interplays between the associated conditions (CVD vs. PD; DM vs. PD; osteoporosis vs. PD) have not been explored yet. The investigators propose to approach this using an integrative in silico method, combining existing diverse biological information including genomic, epigenetic, expression and protein data. To our knowledge, this is the first time that hierarchical levels of integrative precision medicine will be tested for PD vs. CVD/DM/osteoporosis to generate plausible hypotheses and experimental targets.

ELIGIBILITY:
Inclusion Criteria:

* Women who are willing to consent for requesting dental records;
* Outcome 1 - Women who reported periodontal disease diagnosis at any time point up to the 2006 follow up;
* Outcome 1 - Women whose dental records will be retrievable and usable (retrospectively 2 years and prospectively 1 year at the time of report of periodontal disease diagnosis)
* Outcome 2 - Women who are willing to complete and turn-in the WHS 2018 Annual Follow-up Questionnaire with CDC-AAP oral health questions
* Outcome 2 - Women whose dental records will be retrievable and usable (retrospectively 3 years at the time of 2018 Annual Follow-up Questionnaire turn-in)
* The definition of usable dental records consist of but not exclusive to clinical note, complete periodontal charting, and full-mouth radiographs series (FMX) or panoramic, bite-wing radiographs that could derive a PD diagnosis based on the American Academy of Periodontology 1999 definitions.

Exclusion Criteria:

- Women whose dental records are not retrievable or incomplete.

Ages: 45 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants in this protocol are women in the Women's Health Study that agreed to be contacted for follow-up after the clinical trial ended in 2004~2005.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Validity of self-reported periodontal disease | Dental records will be requested retrospectively around the time of questionnaire turned-in that self-reported periodontal disease was reported. The record will be traced back 2 years and prospectively 1 years at the date of report (total 3 years)
  Cronbach's alpha correlation coefficients will be calculated
Correlation of CDC-AAP periodontal condition questions vs. periodontal disease diagnosis | Dental records will be requested retrospectively (3 years) for participants who will return 2018 annual follow-up questionnaire with CDC-AAP questions
  Correlation coefficients will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Benoit, Study Director — Tufts University; Yau-Hua Yu, DDS, DMSc, Principal Investigator — Tufts University School of Dental Medicine
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yu YH, Doucette-Stamm L, Rogus J, Moss K, Zee RYL, Steffensen B, Ridker PM, Buring JE, Offenbacher S, Kornman K, Chasman DI. Family History of MI, Smoking, and Risk of Periodontal Disease. J Dent Res. 2018 Sep;97(10):1106-1113. doi: 10.1177/0022034518782189. Epub 2018 Jun 21. PMID 29928831
- [Result] Shungin D, Haworth S, Divaris K, Agler CS, Kamatani Y, Keun Lee M, Grinde K, Hindy G, Alaraudanjoki V, Pesonen P, Teumer A, Holtfreter B, Sakaue S, Hirata J, Yu YH, Ridker PM, Giulianini F, Chasman DI, Magnusson PKE, Sudo T, Okada Y, Volker U, Kocher T, Anttonen V, Laitala ML, Orho-Melander M, Sofer T, Shaffer JR, Vieira A, Marazita ML, Kubo M, Furuichi Y, North KE, Offenbacher S, Ingelsson E, Franks PW, Timpson NJ, Johansson I. Genome-wide analysis of dental caries and periodontitis combining clinical and self-reported data. Nat Commun. 2019 Jun 24;10(1):2773. doi: 10.1038/s41467-019-10630-1. PMID 31235808